CLINICAL TRIAL: NCT03638921
Title: 35RC17_8826_NEPHROPAIN Phase APRES : Interest of the Equimolar Oxygen Nitride Mixture (MEOPA) in the Treatment of Pain in Patients Presenting to the Emergency Department for Suspected Renal Colic: a Study BEFORE AFTER
Acronym: NEPHROPAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35RC17_8826_NEPHROPAIN Après; 2018-001652-35 (EudraCT Number); 2018/38 (Other: CPP Est I (Dijon))
Record Dates: First submitted 2018-08-07; First posted 2018-08-20 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Renal Colic
MeSH Terms: conditions — Renal Colic | interventions — Meopa

STUDY DESIGN:
Intervention Model Description: MEOPA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEOPA (Experimental): Patients included in the study will receive MEOPA with a high concentration mask (bottle stored for at least 48 hours horizontally) at a minimum flow rate of 10 L / min under supervision of a health care worker after explanation of use to the patient in a quiet environment (box). MEOPA will be administered for a maximum total duration of 20 minutes, continuously or not depending on the needs of the patient, but after a continuous phase at the beginning of treatment of at least 3 minutes.
  Interventions: Drug: MEOPA

INTERVENTIONS:
Drug: MEOPA — Patients included in the study will receive MEOPA with a high concentration mask (bottle stored for at least 48 hours horizontally) at a minimum flow rate of 10 L / min under supervision of a health care worker after explanation of use to the patient in a quiet environment (box). MEOPA will be administered for a maximum total duration of 20 minutes, continuously or not depending on the needs of the patient, but after a continuous phase at the beginning of treatment of at least 3 minutes.

SUMMARY:
MEOPA (Equimolar Oxygen-Nitrogen Protoxide Mix) is a gas used in emergencies for short-term painful acts. It is often very effective with an analgesic, anxiolytic and muscle relaxant action. It is often combined with other analgesic medicines. It has already been proven in emergency medicine for short-term pain and trauma. It seems that it could be used more particularly for pains of medical origin. A study has already proved its effectiveness in the treatment of migraines in emergencies. The first phase of the NEPHROPAIN study began in 2016 after a favorable opinion from the Regional Ethics Committee. NEPHROPAIN phase AVANT was a prospective non-interventional study on the use of analgesic drugs in nephritic colic in emergencies by Dr. Alexandre Tanneau. This study was conducted at the University Hospital of Rennes and included 60 patients admitted to the emergency department for suspected renal colic. It made it possible to recruit the control group of the NEPHROPAIN study. Its main objective was to describe the suspected population of renal colic in Rennes emergencies, to determine NEPHROPAIN's primary endpoint and the number of NEPHROPAIN needed subjects.

ELIGIBILITY:
Inclusion Criteria :

* Age greater than or equal to 18,
* Presenting a suspicion of renal colic, that is to say a pain at the level of a lumbar fossa radiating towards the external genital organs, of rapidly progressive, non-febrile appearance,
* Having given free, informed and written consent,
* Affiliated to the social security system.

Exclusion Criteria :

* Patient in shock of all types, defined here as an acute cardio-circulatory failure with mean arterial pressure less than 65 mm Hg.
* Oxygen saturation below 93% in ambient air,
* With suspicion of pneumothorax,
* Having a history of emphysema and / or COPD (chronic obstructive pulmonary disease),
* Contraindications to the administration of MEOPA: Patients requiring ventilation in pure oxygen; Intracranial hypertension (headache associated with jet vomiting); Any alteration of the state of consciousness, preventing the cooperation of the patient (Glasgow score less than 15); Head trauma; Pneumothorax; Emphysema bubbles; Gas embolism; Diving accident; Abdominal gas distension; Patient who has recently received an ophthalmic gas (SF6, C3F8, C2F6) used in ocular surgery as long as a gas bubble persists inside the eye and at least for a period of 3 months; Known and unsubstituted deficiency of vitamin B12 or folic acid; Neurological abnormalities of recent appearance and unexplained)
* Contraindication to NSAIDs,
* Patient treated in the long course by analgesic stage 3,
* Pregnant or lactating woman,
* Concomitant participation in another research involving the interventional or minimal risk and minimal human person,
* Major persons subject to legal protection (legal safeguards, guardianship, tutorship) and persons deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | 20 minutes
  Pain Ealuation. Score : 0 to 10. Proportion of individuals whose initial pain evaluation (Digital Scale) is divided by at least two to T20.

SECONDARY OUTCOMES:
Analgesics consumption | 0, 20, 60, 240 minutes and through hospitalization completion (an average of a few hours)
  Proportion of individuals who used analgesics between T0 and T20, between T20 and T60, between T60 and T240, and between T240 and at the end of hospitalization.
Adverse effects related to taking analgesics, | through treatment completion, an average of a few hours
NRS average | 0, 20, 60, 240 minutes and through hospitalization completion (an average of a few hours)
  Pain average (digital scale) at T0 (before administration of the first analgesic, MEOPA or other), T20, T60, T240, and at at the end of hospitalization.
  Average of NRS score (pain evaluation, score : 0 to 10).
Hospitalization time | through hospitalizationcompletion, an average of a few hours
  Hospitalization time in emergency

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Paulhet, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No